CLINICAL TRIAL: NCT05327309
Title: Role of Propranolol as Compared to Bleomycin in Management of Hemangioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Ali Raza Chaudhry, Senior Registrar as principal investigator, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 166SZABMU
Record Dates: First submitted 2022-03-12; First posted 2022-04-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hemangioma; Propranolol
Keywords: Infantile Cutaneous hemangioma; Propranolol treatment; Bleomycin treatment; Efficacy
MeSH Terms: conditions — Hemangioma | interventions — Bleomycin; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Active Comparator): propranolol with a mean dose of 2mg/kg/day in 2 divided doses for a period of 6 months
  Interventions: Drug: Bleomycin
- Bleomycin (Experimental): Bleomycin 15mg diluted in 15 ml of Normal Saline along with a dosage of 0.5 mg/kg for a period of 6 months.
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Bleomycin
  Other Names: Propranolol

SUMMARY:
Infantile hemangiomas are widespread vascular tumours having incidence of 10% and most of them involute spontaneously. However, they are known to be located in proximity of vital organs and can have poor cosmetic and functional sequel if left untreated. A wide range of treatment options are available from expectant therapy to radical surgical excision. Propanolol has also been shown to be effective in treating infantile cutaneous hemangiomas. Similarly, anti-metabolite drugs as bleomycin has also shown promising results. Efficacy in terms of reduction in size of both treatments has been scarcely studied especially in Pakistan.

OBJECTIVE: To assess the efficacy of oral propranolol and intraleisonal bleomycin in the treatment of infantile cutaneous hemangioma in terms of size regression

DETAILED DESCRIPTION:
Material & Methods Study design: Randomised controlled trial Place of study: This is study was conducted in the department of paediatric surgery, children hospital, Pakistan institute of medical sciences, Islamabad Duration of study: 24 months

Number of patients:

Using the WHO sample size calculator with following statistical assumptions Confidence interval = 90% Alpha errors = 5% Anticipated population proportion in Group A = 85%9 Anticipated population proportion in Group B = 62.5%9 Sample size will be 45 cases in each study group. Total number of 90 cases will be required in this study Sampling technique: Probability sampling technique Sélection criteria Inclusion criteria

1. 6 month to 12 yr. of age presenting with infantile hemangioma anywhere on body 2. Both sex included 3. Previously not treated Exclusion criteria On the basis of history and clinical assessment;

1. Patients with previous treatment of hemangioma.
2. Patients who will be lost to follow up
3. Patients who refused to be enrolled in this study
4. Patients who experienced hypersensitivity to propranolol/Bleomycin during treatment or had previous known allergy to the drugs.
5. Patients who had diagnosed Cardiac disease such as heart failure or AV block.
6. Patients with diagnosed Pulmonary disease such as asthma or bronchiolitis.
7. History of impaired renal or liver functions.
8. Diabetes mellitus Collection procedure After approval of synopsis, researcher collected data after taking permission from hospital Ethical Committee. Patients were entertained through outdoor department. Patient was explained about the whole procedure. Brief history and clinical examination and investigations were recorded on a Performa. The patients who were diagnosed cases of any cardiac, pulmonary, renal or hepatic diseases were excluded from study based on history. Diagnosis was established on clinical grounds and Doppler ultrasonography of the hemangioma were done to confirm the diagnosis if needed. Size of hemangioma taken and any skin changes were noted.

Patients were explained about the whole treatment and informed written consent taken.

Number of patients: It was conducted on 90 patients that were divided in equal number to two groups randomly by lottery system.

Group A: Included those who had to be managed with oral propranolol. Group B: included those who had to be managed with intralesional injection bleomycin.

The patients were seen in OPD and followed up in OPD. Patients were randomly divided into two non biased groups. One group i.e. Group A received propranolol with a mean dose of 2mg/kg/day in 2 divided doses for a period of 6 months.

Group B consisted of those who received Bleomycin 15mg diluted in 15 ml of 2% plain lidocaine along with a dosage of 0.5 mg/kg for a period of 6 months. The dose of lidocaine was 3mg/kg. It was injected intralesionaly using a syringe and a 27-gauge. Where needed, a pressure dressing was applied for 24 hours. A total of 6 injections were administered and the interval between injections was 2-4 weeks. The patients were admitted for 24 hrs in ward after General Anesthesia (GA) whereas, if GA was not given patient was monitored in day care. Dosage of bleomycin and nature of anaesthesia (i.e., general anaesthetic, local anaesthetic with or without sedation) were prospectively recorded for every patient and session. Vitals were checked in first 24hr period in both groups and noted. Those patient who exhibited any signs of hypersensitivity during and after administration were also left out.

Follow up were done weekly for 1 month in both groups to see changes in size and skin in both groups. After that the follow up was on monthly basis till 6 months. In each visit patients had full clinical examination including pulse and blood pressure with recording of dimensions of the hemangioma based on direct measurement (in centimetres and length, width, height measurement).Small hemangiomas were measured using vernier calliper and others with measuring scale.

Data was collected on follow up for both groups to confirm regression in size of hemangiomas and complications were noted. Single observer (resident pediatrician) saw the patients in each follow up and final outcome measured at 6th month. All this data was recorded on a Performa from 1st month to 6th month on monthly basis.

Statically analysis Data was analyzed by using statistical package for social sciences (SPSS) version 23.0. Mean and standard deviation was calculated for qualitative variables like age, size at the baseline and at the follow up visit up till 6 month.

Frequency and percentages were presented for qualitative data (sex, efficacy in terms of size of hemangioma). Chi square test was applied to compare efficacy of hemangioma in both groups at each visit. A P value < 0.05 was considered statistically significant. Effect modifiers like age, gender, duration and size of hemangioma were controlled by stratification.

ELIGIBILITY:
Inclusion Criteria:

* 1. 6 month to 12 yr. of age presenting with infantile hemangioma anywhere on body 2. Both sex included 3. Previously not treated

Exclusion Criteria:

On the basis of history and clinical assessment;

1. Patients with previous treatment of hemangioma.
2. Patients who will be lost to follow up
3. Patients who refused to be enrolled in this study
4. Patients who experienced hypersensitivity to propranolol/Bleomycin during treatment or had previous known allergy to the drugs.
5. Patients who had diagnosed Cardiac disease such as heart failure or AV block.
6. Patients with diagnosed Pulmonary disease such as asthma or bronchiolitis.
7. History of impaired renal or liver functions.
8. Diabetes mellitus

   -

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Size change | 02 years
  Size change:
  It is defined as change in size at three or six months compared to baseline size of hemangioma and represented in terms of percentage.
  Percentage size change = Size of hemangioma at 3 or 6 months x 100 Initial Size
  Left over Signs after treatment:
  defined as development of scar, hyperpigmentation or change in texture of skin at the location where hemangioma was previously present.
  Efficacy:
  The efficacy of propranolol and bleomycin will be evaluated for change in the size of the lesion, change in the colour of the lesion, epithelialisation in case of ulceration, complications following therapy, and signs of relapse after therapy. The outcome based on change in size will be graded as follows:
  I Complete involution, implying greater than 90percent response. II Response of change in size of 75 to 90percent III Response of change in size of 50 to 75percent. IV Response of change in size of 25 to 50 percent
Size Regression Efficacy Complications: | 2 years
  Objective To evaluate the efficacy of oral propranolol as compared to intralesional Bleomycin in management of cutaneous infantile hemangioma in terms of size change.
  Operational Definition
  Infantile Hemangiomas:
  These are vascular neoplasms which are lesions characterized by abnormal proliferation of endothelial cells and aberrant blood vessel architecture which proliferate after birth and are diagnosed clinically as cherry red vascular lesions.
  Complications:
  Propranolol:
  The known complications which could be present in group taking propranolol were hypotension, pulmonary symptoms as wheeze and precipitation of asthma and hypoglycemia. These findings were carefully looked for in the group taking propranolol.
  Bleomycin:
  The known complications which could be present in group taking bleomycin were Pulmonary symptoms as shortness of breath, bleeding and ulceration of lesions. These symptoms and signs were monitored in patients who were give intra-lesional bleomycin.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Its available

REFERENCES:
- [Result] Thayal PK, Bhandari PS, Sarin YK. Comparison of efficacy of intralesional bleomycin and oral propanolol in management of hemangiomas. Plast Reconstr Surg. 2012 Apr;129(4):733e-735e. doi: 10.1097/PRS.0b013e318245e739. No abstract available. PMID 22456397
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/22456397/
- Available data/document: Individual Participant Data Set — http://pubmed.ncbi.nlm.nih.gov/22456397/